CLINICAL TRIAL: NCT06988241
Title: Efficacy of Positional Release Muscles for Neck Pain During Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Norhan Hassan Elsayed, Physical Therapist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFSIRB200-439
Record Dates: First submitted 2025-05-17; First posted 2025-05-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional Release (Experimental): Positional Release For upper trapezius + Posture correction advices during lactation + posture correction exercises
  Interventions: Other: positional release; Other: Posture correction
- Posture correction (Other): Posture correction advices during lactation + posture correction exercises
  Interventions: Other: Posture correction

INTERVENTIONS:
Other: positional release — All participants in group (A) will receive the same program of group B added to positional release . In order to make the positional release , the therapist will pick up the trigger points by palpation in the upper trapezius muscle by pincer palpation method and distinguished with dots on the skin. Participants will be made supine lying and relaxed by maintaining the cervical spine in a neutral position. Lateral flexion of subject's head toward the side of a tender point, the therapist grasps the subject's forearm and abducts shoulder to approximately 90° and adds slight flexion or extension to fine-tune.The most comfortable position achieved will be held for 90 seconds and after that passive return of the body part to an anatomically neutral position will be maintained for 5 minutes. All participants will be treated three times per week for 4 consecutive weeks and will be instructed to maintain their normal activities while avoiding any undue stress to the neck.
  Other Names: strain counter strain
  Arms: Positional Release
Other: Posture correction — Posture correction advices during lactation + posture correction exercises

SUMMARY:
Purpose of the study: To determine the efficacy of neck muscles positional release for Neck Pain during lactation.Methods:Fifty patient with postpartum neck pain will be recruited. Patients will be randomly assigned into two groups, group A and group B . Patients in both groups will receive posture correction advices during lactation and posture correction exercises but group A will receive additional positional release for upper trapezius. All patients will be evaluated for Pressure pain threshold (PPT) of upper trapezius by algometry, neck disability using Arabic version of neck disability index, pain intensity using 11-numerical rating scale.

DETAILED DESCRIPTION:
Treatment procedure Both groups will receive posture education advices during lactation and Posture correction exercise program which will include Strengthening Exercise Program and Spinal Stretches.Spinal stretches were also included .In the intervention program mothers who underwent normal delivery were advised to start home based exercise program after 5 weeks and the caesarean mothers after 2 months of delivery Group (A): will receive Positional release of neck muscles in addition to Posture correction.Positional release technique For deactivation of Trigger Points (TrPs) and decrease spasm Manual approaches. [PRT] was developed by Lawrence H. PRT is a method in which muscles are placed in a position of greatest comfort, and this causes normalization of muscle hypertonicity and fascial tension. Also, it decreases joint hypomobility, increases circulation, followed by a reduction in swelling, decreased pain, and increase muscle strength. The practical section of the study will be undertaken in 4 weeks (3 sessions a week). Measurement will be taken before the start of treatment program then after the end of 4 weeks treatment program.

ELIGIBILITY:
Inclusion Criteria:

* lactating mothers.
* Age between 25-35 years old.
* six weeks to one year after childbirth.
* at least a moderate level of education.

Exclusion Criteria:

* Mothers were excluded if they had facet joint, neurological, or cardio vascular and respiratory conditions.
* History of breast cancer.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Intensity of neck pain | baseline and four weeks
  Neck pain intensity will be measured by 11- numerical rating scale.Primary outcome updated to pain intensity to better reflect the study objective.

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | baseline and four weeks
  Pressure pain threshold (PPT) of upper trapezius will be measured by digital pressure algometer.
functional status related to neck disability | baseline and four weeks
  Functional status related to neck disability will be measured by Arabic version of Neck

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy kafr Elsheikh university, KafrElSheikh, kafrElsheikh, Egypt